CLINICAL TRIAL: NCT03782233
Title: Effect to Gastrointestinal Barrier Function During Laparoscopic Gastrectomy With Deep vs Moderate Neuromuscular Blockade.
Brief Title: Study on the Level of Neuromuscular Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: He Huang
Record Dates: First submitted 2018-12-11; First posted 2018-12-20 (Actual); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Neuromuscular Blockade
Keywords: Neuromuscular Blockade; Gastrointestinal Barrier Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep neuromuscular blockade group (Group D) (Experimental): Patients undergoing elective laparoscopic surgery for gastrectomy will be randomized to receive deep neuromuscular blockade (post-tetanic count = 1-2) using high dose rocuronium.
  Interventions: Drug: A continuous intravenous infusion of 0.5-0.6 mg/kg/h Rocuronium Bromide Intravenous Solution (50 Mg/5 mL) to keep the target neuromuscular blockade (PTC = 1-2).
- moderate neuromuscular blockade group (Group M) (Other): Patients undergoing elective laparoscopic surgery for gastrectomy will be randomized to receive moderate neuromuscular blockade (train-of-four count = 1-2) using moderate dose rocuronium.
  Interventions: Drug: A continuous intravenous infusion of 0.2-0.3 mg/kg/h Rocuronium Bromide Intravenous Solution (50 Mg/5 mL) to keep the target neuromuscular blockade (TOF = 1-2).

INTERVENTIONS:
Drug: A continuous intravenous infusion of 0.5-0.6 mg/kg/h Rocuronium Bromide Intravenous Solution (50 Mg/5 mL) to keep the target neuromuscular blockade (PTC = 1-2). — 50 patients undergoing laparoscopic gastrectomy surgery will be allocated to group D. A continuous intravenous infusion of 0.5-0.6 mg/kg/h rocuronium to keep the target neuromuscular blockade (PTC = 1-2).
  Arms: deep neuromuscular blockade group (Group D)
Drug: A continuous intravenous infusion of 0.2-0.3 mg/kg/h Rocuronium Bromide Intravenous Solution (50 Mg/5 mL) to keep the target neuromuscular blockade (TOF = 1-2). — 33 patients undergoing laparoscopic gastrectomy surgery will be allocated to group M. A continuous intravenous infusion of 0.2-0.3 mg/kg/h rocuronium to keep the target neuromuscular blockade (TOF = 1-2).
  Arms: moderate neuromuscular blockade group (Group M)

SUMMARY:
On the basis of moderate pneumoperitoneum pressure(10 mmHg), this study evaluates the effect of different level of neuromuscular blockade to gastrointestinal barrier function during laparoscopic gastrectomy. 83 patients are randomized to 2 arms ,The patients in deep neuromuscular blockade group（group D, PTC=1-2）will receive high dose rocuronium (0.5-0.6 mg/kg/h) ;While the patients in moderate neuromuscular blockade group（group M, TOF=1-2）will receive moderate dose rocuronium (0.2-0.3 mg/kg/h)

ELIGIBILITY:
Inclusion Criteria:

1. Age:40-80;
2. BMI < 30kg/m2；
3. ASA classification:Ⅰ-Ⅲ；
4. Undergoing elective laparoscopic gastrectomy.

Exclusion Criteria:

1. Preoperative history of inflammatory intestinal diseases, intestinal flora disorders, obstructive jaundice, intestinal obstruction, irritable bowel syndrome and other digestive diseases;
2. Severe heart, lung, liver, kidney, brain and other diseases;
3. Serious infection, pancreatitis, burns, trauma, need a large dose, long-term use of antibiotics before the operation;
4. A history of abdominal surgery;
5. Combined with gravis myasthenia, serious electrolyte disorders or neuromuscular diseases.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep Neuromuscular Blockade（Group D）: 50 patients undergoing laparoscopic gastrectomy surgery will be allocated to group D. A continuous intravenous infusion of 0.6 mg/kg/h rocuronium to keep the target neuromuscular blockade (PTC = 1-2).
- Moderate Neuromuscular Blockade (Group M): 33 patients undergoing laparoscopic gastrectomy surgery will be allocated to group M. A continuous intravenous infusion of 0.2 mg/kg/h rocuronium to keep the target neuromuscular blockade (TOF = 1-2).
Period: Overall Study
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Started | 50 | 33
Completed | 46 | 31
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M) | Total
Number analyzed (Participants) | 46 | 31 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.8) | 60.0 (8.1) | 60.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 29 | 22 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 46 | 31 | 77
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (2.8) | 24.3 (2.7) | 23.92 (2.76)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of D-lactic Acid Before the Surgery
Description: The level of D-lactic acid can indicate the damage to the gastrointestinal barrier .
Time Frame: 1 day before the surgery
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
ng/ml | 1100.4 (156.6) | 1087.8 (146.0)

2. Primary Outcome: Plasma Concentration of Diamine Oxidase (DAO) Before the Surgery
Description: The level of DAO can indicate the damage to the gastrointestinal barrier .
Time Frame: 1 day Before the Surgery
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
U/L | 15.5 (3.0) | 16.4 (3.6)

3. Primary Outcome: Total Number of Operational Taxonomic Units (OUTs) of Intestinal Microbiota
Description: Intestinal microbiota was analyzed by 16S rRNA sequencing. To be specific, first, DNA was extracted and quantified. Bacterial 16S rRNA genes of the V3-V4 region were amplified from extracted DNA using the barcoded primers (5'- CCTACGGRRBGCASCAGKVRVGAAT-3') and (5'- GGACTACNVGGGTWTCTAATCC-3'). PCR reactions were performed and the PCR mixture applied to the PCR amplifier. Then, the PCR products were checked for size and specificity by agarose gel electrophoresis and purified. Finally, high-throughput sequencing was performed using the Illumina MiSeq platform.
  The raw reads were filtered to remove low quality sequences and the filtered data were further merged into tags by FLASH(Version 1.2.7). Then the Uchime algorithm in Usearch software was applied to remove chimeric tags. Resulting tags for each sample were clustered into operational taxonomic units(OTUs) at the level of 97% similarity.
  Higher values represent a more abundant amount of bacteria in gut.
Time Frame: the first time of defecation after operation
Population: There were only 8 patients in group D and 5 patients in group M defecating before discharged from hospital.
Measure: Number; unit: units
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 8 | 5
units | 1695 | 1287

4. Primary Outcome: Postoperative Exhaust Time
Description: It's a regular measurement to evaluate the function of gastrointestinal tract . It is calculated from the end of the operation to the time of exhaust.
Time Frame: It is calculated from the end of the operation to the time of exhaust.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
hour | 58.9 (15.9) | 70.5 (26.6)

5. Primary Outcome: Plasma Concentration of D-lactic Acid 24 h After the Surgery
Description: The level of D-lactic acid can indicate the damage to the gastrointestinal barrier .
Time Frame: 24 h after the surgery
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
ng/ml | 1230.7 (138.4) | 1297.5 (147.8)

6. Primary Outcome: Plasma Concentration of Diamine Oxidase (DAO) 24 h After the Surgery
Description: The level of DAO can indicate the damage to the gastrointestinal barrier .
Time Frame: 24 h after the Surgery
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
U/L | 18.1 (3.3) | 26.5 (4.7)

7. Primary Outcome: Relative Abundance of Intestinal Microbiota
Description: Intestinal microbiota is one of the factors related to the recovery of intestinal function. It can be analyzed by 16S rRNA sequencing of the postoperative feces.
Time Frame: the first time of defecation after operation
Population: There were 8 patients group D and 5 patients in group M defecating before being discharged from the hospital.
Measure: Median (Standard Deviation); unit: percentage of all intestinal microbiota
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 8 | 5
percentage of all intestinal microbiota
  Class-Deltaproteobacteria | 0.0010483424321 (0.00) | 0.0010483424321 (0.00)
  Class-Flavobacteriia | 0 (0) | 0.000019780046 (0)
  Order-Desulfovibrionales | 0.0081493789065 (0) | 0.0010483424321 (0)
  Order-Flavobacteriales | 0 (0) | 0.00003956 (0)
  Family-[Tissierellaceae] | 0.0021362449560 (0) | 0.0001186802753 (0)
  Family-Fusobacteriaceae | 0.0005340612390 (0) | 0.0196020254767 (0)
  Family-Desulfovibrionaceae | 0.0081493789065 (0) | 0.0010285623862 (0)
  Family-[Weeksellaceae] | 0 (0) | 0.000019780046 (0)
  Genus-Blautia | 0.0097021125088 (0) | 0.0024725057362 (0)
  Genus-Dialister | 0.0002175805047 (0) | 0.0042724899121 (0)
  Genus-Collinsella | 0.0024329456444 (0) | 0 (0)
  Genus-Fusobacterium | 0.0005340612390 (0) | 0.0196020254767 (0)
  Genus-Bilophila | 0.0050636917477 (0) | 0.0010087823403 (0)
  Genus-Aggregatibacter | 0 (0) | 0.0007120816520 (0)
  Genus-Megasphaera | 0.000059340138 (0) | 0.0019780045889 (0)
  Genus-Neisseria | 0 (0) | 0.000019780046 (0)
  Genus-Selenomonas | 0 (0) | 0.000039560092 (0)
  Genus-Roseburia | 0.000019780046 (0) | 0 (0)
  Genus-TG5 | 0 (0) | 0.000019780045 (0)

8. Primary Outcome: 16s rRNA Sequencing of Postoperative Feces
Description: Alpha and Beta diversity; relative abundance of gut microbiota. Alpha diversity includes Chao 1 index, Shannon index, and Simpson index. A higher value of Chao 1 index corresponds to more abundant number of microbiota. A higher value of Shannon index corresponds to more abundance. And A higher value of Simpson index corresponds to less diversity.
  Bata diversity was assessed by PCoA analysis. A three dimensional scatter plot was presented to visualize the similarities and differences between the two groups.
Time Frame: the first time of defecation after operation
Population: There were 8 patients group D and 5 patients in group M defecating before being discharged from the hospital. There are so much basic data about the 16s rRNA sequencing that we can not upload them. The amount of work was formidable. You may contact with me if necessary for all the sequencing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Deep Neuromuscular Blockade Group (Group D) | Moderate Neuromuscular Blockade Group (Group M)
Number analyzed (Participants) | 8 | 5
score on a scale
  alpha diversity - Chao1 | 763.7 (183.7) | 599.3 (164.0)
  alpha diversity - Shannon index | 4.93 (1.0) | 4.15 (0.9)
  alpha diversity - Simpson index | 0.9 (0.07) | 0.83 (0.1)

9. Secondary Outcome: Duration of Surgery
Description: Time from the first dose of anesthetic to the end of the surgery
Time Frame: From the first dose of anesthetic to the end of the surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
minutes | 155.0 (34.2) | 174.6 (34.9)

10. Secondary Outcome: Surgical Condition Scores Rated by Surgeons
Description: evaluation of the surgical condition by 5 point scale: 5 points: optimal; 4 points: good; 3 points: acceptable; 2 points: poor; 1 point: extremely poor.
Time Frame: During operation, within 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
Participants
  1 point | 0 | 1
  2 points | 0 | 4
  3 points | 3 | 16
  4 points | 9 | 7
  5 points | 34 | 3

11. Secondary Outcome: Duration of CO2 Pneumoperitoneum
Description: Time from the beginning to the end of CO2 pneumoperitoneum
Time Frame: from the beginning to the end of CO2 pneumoperitoneum
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
minute | 132.3 (31.2) | 147.0 (34.8)

12. Secondary Outcome: Duration of Postoperative Hospital Stay
Description: Duration from the day of surgery to the day the patient discharged from the hospital
Time Frame: from the end of surgery to the time of being discharged from hospital
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
days | 9.2 (4.0) | 9.1 (5.1)

13. Secondary Outcome: Postoperative VAS (12 h After Surgery, Rest State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 12 h after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 2.2 (1.4) | 2.1 (1.4)

14. Secondary Outcome: Postoperative VAS (12 h After Surgery, Active State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 12 h after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 3.6 (1.6) | 3.8 (1.4)

15. Secondary Outcome: Postoperative VAS (24 h After Surgery, Rest State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 24 h after surgery
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
points | 1.3 (1.0) | 1.5 (1.2)

16. Secondary Outcome: Postoperative VAS (24 h After Surgery, Active State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 24 h after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 2.7 (1.3) | 3.1 (1.4)

17. Secondary Outcome: Postoperative VAS (48 h After Surgery, Rest State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 48 h after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 0.4 (0.8) | 0.7 (1.0)

18. Secondary Outcome: Postoperative VAS (48 h After Surgery, Active State)
Description: VAS pain score: 0 - completely painless, 10 - unbearable pain.
Time Frame: 48 h after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 1.5 (1.1) | 1.5 (1.1)

19. Secondary Outcome: Surgical Condition Scores Rated by Surgeons (Average Scores)
Description: as for outcome 10
Time Frame: during surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
Number analyzed (Participants) | 46 | 31
units on a scale | 4.6 (0.6) | 3.2 (0.9)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 weeks
Description: Our definitions are consistent with the clinicaltrials.gov.
Arm/Group | Deep Neuromuscular Blockade（Group D） | Moderate Neuromuscular Blockade (Group M)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT03782233/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03782233/ICF_001.pdf